CLINICAL TRIAL: NCT06515223
Title: Improving Pelvic Rehabilitation Using Epidural Stimulation After Spinal Cord Injury
Acronym: ImPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301613
Record Dates: First submitted 2024-07-01; First posted 2024-07-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries; Neuromodulation; Neurogenic Bladder; Neurogenic Bowel; Neurogenic Detrusor Overactivity
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Neurogenic Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Implantation of Epidural Spinal Cord Stimulation to target bladder and bowel function. Applied in combination with Pelvic Floor Muscle Training.
  Interventions: Device: Epidural Spinal Cord Stimulation

INTERVENTIONS:
Device: Epidural Spinal Cord Stimulation — Epidural Spinal Cord Stimulation Mapping and Pelvic Floor Muscle Training

SUMMARY:
The investigators will recruit up to 20 volunteers with chronic, supra-sacral SCI. Following screening, eligible participants will enter 'Phase I', they will complete baseline outcome measures and then have the epidural spinal cord stimulator (eSCS) implanted with either percutaneous or paddle electrodes. Preoperative and intraoperative testing will determine exact location of electrodes.

Mapping and optimisation of stimulation parameters will be performed simultaneously with urodynamic investigations of bladder function, and anorectal physiology investigations of bowel function. The acute effects of eSCS to suppress bladder overactivity, facilitate voiding, prevent unwanted reflex sphincter activity, and pelvic floor function will guide development of eSCS programmes for use at home.

In 'Phase II', participants will use eSCS at home for 12-weeks. Participants will also be taught how to perform bladder and pelvic floor muscle training (PFMT) in combination with eSCS.

Outcome measures assessing bladder, bowel, sexual function, quality of life, motor function and spasticity will be captured prior to and following the 12-week intervention, and at 3 and 6 month follow up.

DETAILED DESCRIPTION:
Screening:

Following confirmation that participants meet the eligibility criteria, they will undergo extensive screening, to confirm their suitability for eSCS implantation. They will meet with multidisciplinary team members, to ensure they are fully educated about the potential risks, and to manage their expectations of outcomes. They will undergo a urodynamics assessment, following standard protocol. If they have neurogenic detrusor overactivity (NDO), and are responsive to dorsal genital nerve stimulation to supress NDO they will progress to have an MRI.

Phase I:

Baseline measurements will be completed as outlined in 'outcome measures'. Participants will undergo implantation of a Senza implantable pulse generator (Nevro Corp., CA, USA), which is MRI-conditional and multi-programmable, with Surpass Surgical or Percutaneous leads (Nevro Corp., CA, USA). The device will be implanted under the skin either at the abdomen, superior to iliac crest, or buttocks.

Participants will attend three mapping sessions to determine effective stimulation sites and parameters for the lower limbs, bladder, bowel and pelvic floor muscles. An optional cardiovascular mapping session will also be offered. The mapping sessions will generate several eSCS programmes for participants to use at home, which target specific effects: supression of NDO, facilitation of voiding, bowel management, and pelvic floor muscle activation.

Participants will have a pelvic floor examination, and be taught a pelvic floor muscle training programme to complete at home. They will be educated on how to use the above programmes as part of their daily routine.

Phase II:

For the following 12-weeks participants will use their eSCS programmes and complete daily PFMT. At week 3, 6 and 9, they will be invited to attend a face to face pelvic floor clinic, to review their programme and progress their exercises as indicated. Participants will be called once a week by a member of the research team to check how the participant is managing with their device/programmes, identify any issues, and have any questions answered. They will be asked to complete a 3-day bladder diary and up to 14-day bowel diary during this period.

Participants will repeat baseline measures (with urodynamics, anorectal physiology and global perception of improvement measure) at the end of the 12-week home trial.

Participants will be offered for their eSCS device to be explanted or they can continue with this in situ. They will have time to consider this and discuss this with the clinical care team and researchers. Irrespective of decision, with participants consent, the investigators will continue to follow them up 3, and 6 months later.

If participants keep the SCS device following the 12-week home trial, the repeat bladder and bowel diary assessments will be captured during a period of 2-weeks without stimulation. They will then be able to proceed with using this device as normal.

All participants will be invited to take part in an interview to discuss their participation in the trial, and their decision to either keep or remove the SCS device. This will be audio recorded which will be destroyed once transformed into a written script.

Participants will return to RNOH Stanmore to complete re-assessment of outcomes at 3 and 6 months.

At the end of the study, participants will be offered for their eSCS device to be explanted or they can continue with this in situ, with ongoing support from The London Spinal Cord Injury Centre team/service.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury (supra-sacral)
* AIS A-D
* >18 years;
* SCI sustained >12 months ago;
* Neurogenic detrusor overactivity (NDO) confirmed on urodynamics;
* Responsive to dorsal genital nerve stimulation
* Willing and able to provide informed consent
* Stable medical, physical and psychological condition as considered by the investigators
* Able to understand and interact with the study team in English
* Sufficient upper limb function to operate the device
* Suitably optimised bladder and bowel routine

Exclusion Criteria:

* Transected cord or SCI related to a neurodegenerative disease
* Any device or metal work in situ that would exclude the patient from having eSCS implanted
* Intra-detrusor botulinum toxin injections within the last 6 months
* Previous surgical intervention on bladder sphincters
* Any diseases and conditions that would exclude the patient from eSCS and/or surgery, for example, degenerative spinal pathology, syrinx and/or tumor.
* Recurrent urinary tract infection refractory to antibiotics
* Women who are pregnant or intending to become pregnant (pregnancy test obligatory for woman of childbearing potential) or breast feeding, or lack of safe contraception for women of childbearing capacity.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders or dementia of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Maximum Cystometric Capacity (bladder capacity) from baseline (week 1) to post intervention (week 16) and follow up (week 28, week 40) | Week 1, 16, 28 and 40
  During standard cystometry (retrograde filling of the bladder), maximum cystometric capacity will be defined as the volume emptied from the bladder after each fill.

SECONDARY OUTCOMES:
Maximum Detrusor Pressure | Week 1, 16, 28 and 40
  Maximum recorded detrusor pressure during standard cystometry (retrograde filling of the bladder).
Rectal and Anal Pressure during Push Manoeuvre | Week 3, 16, 28 and 40
  During standard anorectal physiology, London protocol.
3 day bladder diary | Week 3, 12, 16, 28 and 40
  Bladder diary will be completed on clinically used bladder diaries. Participants will record voided volumes, urinary incontinence episodes and daily spasticity for 3 days. This will involve measuring the volume voided each time they urinate over the three days, using provided measuring equipment.
Up to 14 day bowel diary | Week 3, 12, 16, 28 and 40
  Bowel diary will be completed on clinically used bowel diaries. Participants will record type of stool and amount, bowel incontience, bowel management e.g laxatives, use of manual evacuation.
Questionnaire - Neurogenic Bladder Symptom Score (NBSS) | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Scored as 3 subscales - incontinence, score 0-12 (higher score, more severe symptoms), storage and voiding, score 0-9 (higher score, more severe symptoms), and consequences, score 0-7 (higher score, more severe symptoms).
Questionnaire - Urinary Symptom Profile questionnaire | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Scored as 3 subscales - stress urinary incontinence, score 0-9 (higher score, more severe symptoms), overactive bladder, score 0-21 (higher score, more severe symptoms), and low stream, score 0-9 (higher score, more severe symptoms).
Questionnaire - Neurogenic Bowel Dysfunction Score (NBDS) | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Total score, from 0-47 (higher score, more severe symptoms). General satisfaction score 0-10, 0=total dissatisfaction, 10=perfect satisfaction.
Questionnaire - EQ-5D-5L Quality of Life questionnaire | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Scored from 1-5 for each health state (1 indicates no problem, 5 indicates unable to/extreme problems). VAS is scored 0-100 (0 refers to 'the worst health you can imagine', 100 refers to 'the best health you can imagine').
Questionnaire - ISCOS Lower Urinary Tract Dysfunction Dataset (LUTDD) | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Not a scored questionnaire - obtains information about LUT function.
Questionnaire - The International Index of Erectile Function (IIEF) or The Female Sexual Function Index (FSFI) | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  IIEF:
  Questions scored 0-5 or 1-5, (higher score, more severe symptoms). Total score, minimum 6, maximum 75 (higher score, more severe symptoms).
  FSFI:
  Questions scored 0-5 or 1-5, (higher score, more severe symptoms). Total score, minimum 2, maximum 36 (higher score, more severe symptoms).
Questionnaire - Penn Spasm Frequency Scale | Week 2, 16, 28 and 40
  Participants will be asked to complete the questionnaire in a private room at RNOH Stanmore.
  Frequency score 0-4, (higher score, more severe symptoms). Severity score 1-3, (higher score, more severe symptoms).
The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Week 2, 16, 28 and 40
  Sensory and motor examination to determine classification of SCI, level of injury and completeness of the injury.
Colonic Transit Assessment | Week 2, 12 and 40
  A colonic transit study is a test that shows how quickly food passes through the digestive system. Participants will swallow tablets on three consecutive days. On the fourth day, they will have an x-ray.
Microbiome Testing | Week 2, 16 and 40
  Poo sample will be collected by participant, and bacteria present analysed.

CONTACTS AND LOCATIONS:
Overall Officials: David Baxter, MD, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No